CLINICAL TRIAL: NCT05748002
Title: Prediction for Abnormal Topography Corneas Using New Biomechanical Parameter - Biomechanical Stable Index
Brief Title: Evaluation of Morphology Abnormal Cornea Stability With Corneal Biomechanical
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023002
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Keratoconus, Stable
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- stable group
  Interventions: Other: Pentacam and Corvis ST
- subclinical keratoconus
  Interventions: Other: Pentacam and Corvis ST
- normal group
  Interventions: Other: Pentacam and Corvis ST
- follow up group
  Interventions: Other: Pentacam and Corvis ST

INTERVENTIONS:
Other: Pentacam and Corvis ST — morphological and biomechanical parameters of corneal were obtain by Pentacam and Corvis ST

SUMMARY:
To evaluate the corneal biomechanical properties of stable eyes with abnormal morphology, and introduce a biomechanical stable index to evaluate the stability of the eyes with abnormal morphology at the first diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Best corrected visual acuity (BCVA) ≥ 20/20;
2. No other eye diseases except myopia and astigmatism;
3. The cornea was transparent, and there was no cloud or pannus;
4. No clinical manifestation of keratoconus（Corneal stromal thinning, Cone-shaped anterior protrusions, Fleischers ring, Vogts striae, Epithelial or subepithelial scarring） Exclusion Criteria:1) corneal disease;

2) ocular trauma; 3) Patients were required to stop wearing soft contact lenses for at least 2 weeks and rigid contact lenses for at least 4 weeks before examination; 4) Pregnant and lactating women;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients premedicated for refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
stable | one year
  No alterations in morphological(Pentacam parameters, BAD<0.42, TCT<10μm) and biomechanical(Corvis ST, parametersCBI<0.2, SPA1<10) parameters between the first and last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided